CLINICAL TRIAL: NCT03336502
Title: Pharmacokinetics and Safety of Intravenous Posaconazole (MK-5592, POS) in Chinese Subjects at High Risk for Invasive Fungal Infections
Brief Title: Pharmacokinetics and Safety of Intravenous Posaconazole (MK-5592) in Chinese Participants at High Risk for Invasive Fungal Infections (MK-5592-120)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 5592-120; MK-5992-120 (Other: Protocol Number)
Record Dates: First submitted 2017-11-06; First posted 2017-11-08 (Actual); Results first posted 2019-12-19 (Actual); Last update posted 2019-12-19 (Actual); Status verified 2019-12

CONDITIONS: Fungal Infection
MeSH Terms: conditions — Mycoses | interventions — posaconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Posaconazole (Experimental): All participants will receive posaconazole 300 mg intravenous (IV) infusion twice on Day 1 followed by 300 mg IV infusion once daily on Days 2 to 10 (±1). At the discretion of the investigator, participants will received posaconazole 300 mg IV infusion once daily or 200 mg oral suspension three times daily for up to 18 additional days.
  Interventions: Drug: Posaconazole

INTERVENTIONS:
Drug: Posaconazole — Posaconazole 18 mg/mL IV solution; posaconazole 40 mg/mL oral suspension
  Other Names: MK-5592; Noxafil

SUMMARY:
The purpose of this study is to evaluate the pharmacokinetics and safety of posaconazole intravenous solution in Chinese participants at high risk for invasive fungal infections. Neutropenic participants undergoing chemotherapy for acute myelogenous leukemia or myelodysplastic syndromes will be enrolled in the study. The primary hypothesis is to evaluate the pharmacokinetic parameters of intravenous (IV) posaconazole (POS) solution in Chinese participants at high risk of invasive fungal infections and determine the percentage of Chinese participants who reach steady-state concentration averages of POS in blood plasma of 500 ng/ml and higher. Two subgroups were evaluated: Subgroup 1 from serial PK blood draw sampling and Subgroup 2 from sparse limited PK blood draw sampling.

ELIGIBILITY:
Inclusion Criteria:

* Chinese participant
* Female of reproductive potential with a serum of beta human chorionic gonadotropin (β-hCG) level consistent with a nongravid state and agree and/or have their partner use 2 acceptable methods of birth control throughout the study
* Body Mass Index (BMI) >=15 and <=30 kg/m^2
* Have a central line catheter or peripherally central venous catheter in place
* Anticipated or documented prolonged neutropenia and likely to last for at least 7 days due to: a) standard intensive chemotherapy, anthracycline-based or other accepted regimen (excluding any investigational agent) for a new diagnosis of acute myelogenous leukemia (AML); b)chemotherapy for AML in first relapse; or c) therapy for myelodysplastic syndromes in transformation to AML or other diagnoses of secondary AML (therapy related, antecedent hematological disorders) other than chronic myelogenous leukemia in blast crisis
* Free from any clinically significant disease other than the primary hematologic disease that would interfere with administration of study medication or study evaluations
* Able to tolerate central IV solution

Exclusion Criteria:

* Pregnant, intends to become pregnant during the study, or has been nursing
* Mentally or legally incapacitated, has significant emotional problems, or has clinically significant psychiatric disorder over the last 5 years
* Received systemic antifungal therapy (oral, intravenous, or inhaled) within 30 days of study enrollment for reasons other than antifungal prophylaxis
* Known or suspected invasive or systemic fungal infection
* Taken posaconazole within 10 days prior to study enrollment
* Major surgery, donated or lost 1 unit of blood, or participated in another investigational study within 4 weeks prior to the study
* Type 1 hypersensitivity or idiosyncratic reactions to azole agents
* Significant multiple or severe allergies, or has had an anaphylactic reaction or significant intolerability to drugs or food
* Moderate or severe liver dysfunction
* Chronic active hepatitis, cirrhosis, Hepatocellular Carcinoma (HCC), or other hepatic disease caused by a virus
* Previous electrocardiogram with a prolonged QTc interval
* Prior enrollment in this study or other posaconazole studies within 90 days of study entry
* Eastern Cooperative Oncology Group (ECOG) performance status was >2 prior to induction chemotherapy for the underlying disease
* Known or suspected Gilbert's disease.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2017-12-20 (Actual); Primary Completion 2018-11-26 (Actual); Study Completion 2018-11-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (7):
- China (7):
  - Guangdong General Hospital, Guangdong Academy of Medical Science ( Site 0002), Guangzhou, Guangdong
  - The First Affiliated Hospital of Soochow University ( Site 0004), Suzhou, Jiangsu
  - Peking University People's Hospital ( Site 0008), Beijing
  - Peking University Third Hospital ( Site 0009), Beijing
  - Peking Union Medical College Hospital ( Site 0006), Beijing
  - Shanghai General Hospital ( Site 0007), Shanghai
  - Institute of Hematology and Blood Diseases Hosp CAMS&PUMC ( Site 0001), Tianjin

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Wu D, Mi Y, Weng J, Zhuang J, Ke X, Wang C, Liu K, Martinho M, Winchell GA, Zang Y, Xu L. Phase 1b/3 Pharmacokinetics and Safety Study of Intravenous Posaconazole in Adult Asian Participants at High Risk for Invasive Fungal Infections. Adv Ther. 2022 Apr;39(4):1697-1710. doi: 10.1007/s12325-021-02012-1. Epub 2022 Feb 15. PMID 35167031

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 70 participants were randomized and 70 received at least one dose of study drug.
Groups:
- Serial PK (Subgroup 1): Posaconazole (POS) 300 mg intravenous (IV) infusion twice on Day 1 followed by 300 mg IV infusion once daily on Days 2 to 10 (±1). At the discretion of the investigator, participants may have received POS 300 mg IV infusion once daily or 200 mg oral suspension 3 times daily for up to 18 additional days. Serial PK requires full intensive blood sampling for PK measurements
- Sparse PK (Subgroup 2): POS 300 mg intravenous (IV) infusion twice on Day 1 followed by 300 mg IV infusion once daily on Days 2 to 10 (±1). At the discretion of the investigator, participants may have received POS 300 mg IV infusion once daily or 200 mg oral suspension 3 times daily for up to 18 additional days. Sparse PK requires sparse infrequent blood sampling for PK measurements
Period: Overall Study
Arm/Group | Serial PK (Subgroup 1) | Sparse PK (Subgroup 2)
Started (70) | 30 | 40
Completed (57) | 26 | 31
Not Completed | 4 | 9
Not completed — Physician Decision | 0 | 1
Not completed — Prohibited Drugs | 1 | 1
Not completed — Death | 1 | 2
Not completed — Adverse Event | 2 | 5

BASELINE CHARACTERISTICS:
Population: Subgroup 1 - Serial PK group, received at least 10 days of POS, and analyzed for plasma trough determination AND PK parameters Subgroup 2 - Sparse PK group, received at least 10 days of POS, and analyzed for plasma trough determination.
  Both groups received the same dose and drug administration, reflect only different blood sampling schedules.
Groups:
- Total: Total of all reporting groups
Arm/Group | Serial PK (Subgroup 1) | Sparse PK (Subgroup 2) | Total
Number analyzed (Participants) | 30 | 40 | 70
Age, Continuous [Mean (Standard Deviation); unit: Years]
  18 to 70 Years of Age | 39.8 (13.3) | 45.4 (15.1) | 43 (14.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 20 | 34
  Male | 16 | 20 | 36
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 30 | 40 | 70
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 30 | 40 | 70
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Steady State (ss) Average Concentration (Cavg) of Posaconazole of Serial PK (Subgroup 1) on Day 10
Description: Characterization of the pharmacokinetics (PK) parameters of POS determined from plasma samples taken at steady-state after receiving IV administration of 300 mg POS twice a day (BID) on Day 1 and then 300 mg POS QD until at least Day 10. Steady-state Cavg, where Cavg is defined as AUC0-24hr divided by the dosing interval.
  Subgroup 1 - Serial PK, multiple same-day blood draw, performed specifically for determination of PK parameters of Cavg, AUC, Cmin, Cmax, Tmax and Total Body Clearance in addition to plasma trough determination.
  Subgroup 2 - Sparse PK, once a day blood draw, performed for plasma trough determination only.
Time Frame: Serial PK (Subgroup 1) on Day 10 at pre-dose, 1 hr. post start of infusion (SOI), end of infusion (EOI), 15 min. after EOI and 4, 8, 12, 24 hours post SOI
Population: Analysis population includes participants who had serial blood draws on Day 10. Sparse PK (subgroup 2) is not included in this analysis because blood was drawn only once on Day 10 for plasma trough determination.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Serial PK (Subgroup 1) | Sparse PK (Subgroup 2)
Number analyzed (Participants) | 27 | 0
ng/mL | 2986.28 (1074.5) |

2. Primary Outcome: Percentage of Participants With ssCavg ≥500 ng/mL of Serial PK (Subgroup 1) on Day 10
Description: Characterization of the PK parameters of POS determined from plasma samples taken at steady-state after receiving IV administration of 300 mg POS twice a day (BID) on Day 1 and then 300 mg POS QD until at least Day 10. Steady-state Cavg, where Cavg is defined as AUC0-24hr divided by the dosing interval. The percentage of participants with ssCavg ≥500 ng/mL are presented.
  Subgroup 1 - Serial PK, multiple same-day blood draw, performed specifically for determination of PK parameters of Cavg, AUC, Cmin, Cmax, Tmax and Total Body Clearance in addition to plasma trough determination.
  Subgroup 2 - Sparse PK, once a day blood draw, performed for plasma trough determination only.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | Serial PK (Subgroup 1) | Sparse PK (Subgroup 2)
Number analyzed (Participants) | 27 | 0
Percentage of Participants
  Cavg 500 ng/mL to < 2500 ng/mL | 40.7 |
  Cavg 2500 ng/ML to < 3650 ng/mL | 33.3 |
  Cavg 3650 ng/mL or higher | 25.9 |

3. Primary Outcome: Steady-state Area Under the Concentration-time Curve (ssAUC0-24hr) of POS of Serial PK (Subgroup 1) on Day 10
Description: Characterization of the PK parameters of POS determined from plasma samples taken at steady-state after receiving IV administration of 300 mg POS twice a day (BID) on Day 1 and then 300 mg POS QD until at least Day 10. AUC0-24 is defined as area under the plasma concentration-time curve from time 0 extrapolated to 24 hours.
  Subgroup 1 - Serial PK, multiple same-day blood draw, performed specifically for determination of PK parameters of Cavg, AUC, Cmin, Cmax, Tmax and Total Body Clearance in addition to plasma trough determination.
  Subgroup 2 - Sparse PK, once a day blood draw, performed for plasma trough determination only.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | Serial PK (Subgroup 1) | Sparse PK (Subgroup 2)
Number analyzed (Participants) | 27 | 0
hr*ng/mL | 71670.8 (25788.11) |

4. Primary Outcome: Steady State Maximum Concentration (ssCmax) of POS of Serial PK (Subgroup 1) on Day 10
Description: Characterization of the PK parameters of POS determined from plasma samples taken at steady-state after receiving IV administration of 300 mg POS twice a day (BID) on Day 1 and then 300 mg POS QD until at least Day 10. Cmax is defined as the maximum concentration of POS in plasma.
  Subgroup 1 - Serial PK, multiple same-day blood draw, performed specifically for determination of PK parameters of Cavg, AUC, Cmin, Cmax, Tmax and Total Body Clearance in addition to plasma trough determination.
  Subgroup 2 - Sparse PK, once a day blood draw, performed for plasma trough determination only.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Serial PK (Subgroup 1) | Sparse PK (Subgroup 2)
Number analyzed (Participants) | 27 | 0
ng/mL | 4612.22 (1221.68) |

5. Primary Outcome: Steady State Minimum Concentration (ssCmin) of POS of Serial PK (Subgroup 1) on Day 10
Description: Characterization of the PK parameters of POS determined from plasma samples taken at steady-state after receiving IV administration of 300 mg POS twice a day (BID) on Day 1 and then 300 mg POS QD until at least Day 10. Cmin is defined as the minimum concentration of POS in plasma.
  Subgroup 1 - Serial PK, multiple same-day blood draw, performed specifically for determination of PK parameters of Cavg, AUC, Cmin, Cmax, Tmax and Total Body Clearance in addition to plasma trough determination.
  Subgroup 2 - Sparse PK, once a day blood draw, performed for plasma trough determination only.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Serial PK (Subgroup 1) | Sparse PK (Subgroup 2)
Number analyzed (Participants) | 27 | 0
ng/mL | 2311.33 (1119.28) |

6. Primary Outcome: Time to Steady-state Maximum Concentration (ssTmax) of POS of Serial PK (Subgroup 1) on Day 10
Description: Characterization of the PK parameters of POS determined from plasma samples taken at steady-state after receiving IV administration of 300 mg POS twice a day (BID) on Day 1 and then 300 mg POS QD until at least Day 10. Tmax is defined as the time it takes to achieve maximum concentration of POS in plasma.
  Subgroup 1 - Serial PK, multiple same-day blood draw, performed specifically for determination of PK parameters of Cavg, AUC, Cmin, Cmax, Tmax and Total Body Clearance in addition to plasma trough determination.
  Subgroup 2 - Sparse PK, once a day blood draw, performed for plasma trough determination only.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | Serial PK (Subgroup 1) | Sparse PK (Subgroup 2)
Number analyzed (Participants) | 27 | 0
hr | 1.63 (0.23) |

7. Primary Outcome: Total Body Clearance (CL) of POS of Serial PK (Subgroup 1) on Day 10
Description: Characterization of the PK parameters of POS determined from plasma samples taken at steady-state after receiving IV administration of 300 mg POS twice a day (BID) on Day 1 and then 300 mg POS QD until at least Day 10. CL is defined as the time it takes for POS to be completely removed from the body's blood stream.
  Subgroup 1 - Serial PK, multiple same-day blood draw, performed specifically for determination of PK parameters of Cavg, AUC, Cmin, Cmax, Tmax and Total Body Clearance in addition to plasma trough determination.
  Subgroup 2 - Sparse PK, once a day blood draw, performed for plasma trough determination only.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mL/hr
Arm/Group | Serial PK (Subgroup 1) | Sparse PK (Subgroup 2)
Number analyzed (Participants) | 27 | 0
mL/hr | 4767.90 (1805.24) |

8. Primary Outcome: POS Plasma Trough Concentrations in the Serial PK and Sparse PK Subgroups
Description: Pre-dose plasma trough concentrations by study day between serial PK and Sparse PK - where serial PK is defined as multiple serial blood sampling of more than 6 timepoints; and sparse PK is defined as few blood samples taken and single or limited timepoints
Time Frame: Day 3, Day 6, Day 10, Day 15, Day 22, Day 28
Population: All evaluable participants in Subgroup 1 (Serial PK) and Subgroup 2 (Sparse PK) not yet switched to oral suspension.
  Both groups received the same dose and drug administration and reflect only different blood sampling schedules.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Serial PK (Subgroup 1) | Sparse PK (Subgroup 2)
Number analyzed (Participants) | 30 | 40
ng/mL
  Day 3: number analyzed (Participants) | 30 | 38
  Day 3 | 1800.93 (525.20) | 2033 (650.9)
  Day 6: number analyzed (Participants) | 28 | 35
  Day 6 | 2106.07 (764.16) | 2514 (927.5)
  Day 10: number analyzed (Participants) | 27 | 30
  Day 10 | 2473.78 (1247.86) | 2466 (1045)
  Day 15: number analyzed (Participants) | 8 | 11
  Day 15 | 2471.63 (1495.20) | 2680 (1269)
  Day 22: number analyzed (Participants) | 0 | 6
  Day 22 |  | 2603 (1325)
  Day 28: number analyzed (Participants) | 0 | 2
  Day 28 |  | 3180 (1527)

9. Secondary Outcome: Adverse Events (AEs)
Description: Number of participants with one or more AEs where AEs are defined as any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.
Time Frame: Up to 58 days
Population: All participants who received at least one dose of study drug.
Measure: Number; unit: Number of Participants
Groups:
- POS IV (MK-5592): POS 300 mg intravenous (IV) infusion twice on Day 1 followed by 300 mg IV infusion once daily on Days 2 to 10 (±1). At the discretion of the investigator, participants may have received POS 300 mg IV infusion once daily or 200 mg oral suspension 3 times daily for up to 18 additional days.
Arm/Group | POS IV (MK-5592)
Number analyzed (Participants) | 70
Number of Participants | 70

10. Secondary Outcome: Discontinuations Due to an AE
Description: Number of participants discontinued from study medication due to an AE where AEs are defined as any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.
Time Frame: Up to 28 days
Population: All participants who received at least one dose of study drug.
Measure: Number; unit: Participants
Arm/Group | POS IV (MK-5592)
Number analyzed (Participants) | 70
Participants | 9

11. Secondary Outcome: Medically Significant Changes in Clinical Laboratory Results - Lab Values
Description: The number of participants with clinical laboratory values outside of normal range
Time Frame: Up to 28 days
Population: as for outcome 8
Measure: Number; unit: Participants
Arm/Group | Serial PK (Subgroup 1) | Sparse PK (Subgroup 2)
Number analyzed (Participants) | 30 | 40
Participants | 30 | 35

12. Secondary Outcome: Medically Significant Changes in Clinical Laboratory Results - Vital Signs
Description: The number of participants with values of vital signs outside of normal range
Time Frame: Up to 28 days
Population: as for outcome 8
Measure: Number; unit: Participants
Arm/Group | Serial PK (Subgroup 1) | Sparse PK (Subgroup 2)
Number analyzed (Participants) | 30 | 40
Participants | 27 | 31

13. Secondary Outcome: Survival Status
Description: Survival assessment as to whether a participant is alive or dead, included all participants who died - 2 during study treatment, 1 during safety follow-up, 2 during survival follow-up (Day 60 to 70 post dose), and 1 participant who died during serious AE (SAE) follow-up at 97 days after first dose but was beyond the safety and the survival follow-up period
Time Frame: Up to 98 days
Population: All participants who received at least one dose of study drug.
Measure: Number; unit: Participants
Arm/Group | POS IV (MK-5592)
Number analyzed (Participants) | 70
Participants
  Alive | 64
  Dead | 6

14. Secondary Outcome: Participants With Invasive Fungal Infection (IFI)
Description: Number of participants with possible, probable, or proven IFI observed during the whole study period
Time Frame: Up to 28 days
Population: All participants who received at least one dose of study drug.
Measure: Number; unit: Participants
Arm/Group | POS IV (MK-5592)
Number analyzed (Participants) | 70
Participants | 2

ADVERSE EVENTS:
Time Frame: Up to 98 days post first study dose
Description: All participants who received at least one dose of study drug.
Arm/Group | POS IV (MK-5592)
All-Cause Mortality (participants affected / at risk) | 6/70
Serious Adverse Events (participants affected / at risk) | 15/70
Other Adverse Events (participants affected / at risk) | 70/70
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | POS IV (MK-5592) (N=70)
Agranulocytosis (Blood and lymphatic system disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 4 (4)
Cardiac failure (Cardiac disorders) | 2 (2)
Lung infection (Infections and infestations) | 1 (1)
Tuberculosis (Infections and infestations) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Distributive shock (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | POS IV (MK-5592) (N=70)
Anaemia (Blood and lymphatic system disorders) | 33 (64)
Febrile neutropenia (Blood and lymphatic system disorders) | 4 (5)
Leukocytosis (Blood and lymphatic system disorders) | 4 (4)
Leukopenia (Blood and lymphatic system disorders) | 13 (25)
Thrombocytopenia (Blood and lymphatic system disorders) | 10 (17)
Abdominal distension (Gastrointestinal disorders) | 6 (6)
Abdominal pain (Gastrointestinal disorders) | 4 (4)
Abdominal pain upper (Gastrointestinal disorders) | 6 (9)
Constipation (Gastrointestinal disorders) | 18 (21)
Diarrhoea (Gastrointestinal disorders) | 24 (28)
Gingival ulceration (Gastrointestinal disorders) | 6 (6)
Nausea (Gastrointestinal disorders) | 29 (44)
Proctalgia (Gastrointestinal disorders) | 4 (4)
Vomiting (Gastrointestinal disorders) | 22 (33)
Asthenia (General disorders) | 14 (22)
Chest discomfort (General disorders) | 10 (13)
Chest pain (General disorders) | 4 (4)
Oedema peripheral (General disorders) | 6 (7)
Pyrexia (General disorders) | 40 (81)
Gastrointestinal infection (Infections and infestations) | 4 (4)
Lung infection (Infections and infestations) | 12 (12)
Oral infection (Infections and infestations) | 6 (6)
Upper respiratory tract infection (Infections and infestations) | 8 (8)
Alanine aminotransferase increased (Investigations) | 16 (22)
Aspartate aminotransferase increased (Investigations) | 8 (10)
Blood bilirubin increased (Investigations) | 28 (39)
Brain natriuretic peptide increased (Investigations) | 6 (6)
Gamma-glutamyltransferase increased (Investigations) | 4 (4)
Lymphocyte count decreased (Investigations) | 38 (112)
Neutrophil count decreased (Investigations) | 40 (81)
Platelet count decreased (Investigations) | 32 (88)
Weight increased (Investigations) | 9 (10)
White blood cell count decreased (Investigations) | 50 (108)
Decreased appetite (Metabolism and nutrition disorders) | 9 (10)
Hyperglycaemia (Metabolism and nutrition disorders) | 18 (28)
Hyperuricaemia (Metabolism and nutrition disorders) | 5 (5)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 22 (35)
Hypocalcaemia (Metabolism and nutrition disorders) | 17 (32)
Hypokalaemia (Metabolism and nutrition disorders) | 46 (75)
Hyponatraemia (Metabolism and nutrition disorders) | 16 (23)
Hypophosphataemia (Metabolism and nutrition disorders) | 6 (7)
Hypoproteinaemia (Metabolism and nutrition disorders) | 8 (13)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (4)
Dizziness (Nervous system disorders) | 10 (18)
Headache (Nervous system disorders) | 5 (6)
Poor quality sleep (Nervous system disorders) | 4 (8)
Insomnia (Psychiatric disorders) | 4 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 14 (18)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 7 (9)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 8 (10)
Rash (Skin and subcutaneous tissue disorders) | 12 (14)
Hypertension (Vascular disorders) | 5 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission; this confidentiality does not include efficacy and safety results. Sponsor review can be expedited to meet publication timelines.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-07-24): https://cdn.clinicaltrials.gov/large-docs/02/NCT03336502/Prot_SAP_000.pdf